CLINICAL TRIAL: NCT00546442
Title: Effect of Treatment of Insulin Resistance in Patients With Chronic Hepatitis C Genotype 1 Treated With Peginterferon Alfa-2a in Combination With Ribavirin in Current Clinical Practice
Brief Title: Treatment Insulin Resistence in HCV G-1 Patient
Acronym: TRIC-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Valme University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-02446-19
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Chronic Hepatitis C
Keywords: insulin resistance; chronic hepatitis C; genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Placebo of metformine 850-2550 mg/daily for 48 weeks
  Interventions: Other: Placebo of metformine
- 1 (Experimental): Metformine 850-2550 mg/daily for 48 weeks
  Interventions: Drug: Metformine

INTERVENTIONS:
Drug: Metformine — 850-2550 mg/daily for 48 weeks
  Arms: 1
Other: Placebo of metformine — 850-2550 mg/daily for 48 weeks
  Arms: 2

SUMMARY:
To evaluate the effect of treatment of insulin resistance in the response of chronic hepatitis C treatment, mesure as HCV-RNA negative at week 72.

4.3.2 Objetivos secundarios To evaluate the efficacy and safety of treatment with metformine to erradicate the insulin resistance of patients with chornic hepatitis C genotype 1 measure as HOMA-IR < 2.

DETAILED DESCRIPTION:
Differents studies show that infection by virus hepatitis C have a relevant rol in the development of insulin resistance. The insulin resistence is associated with a progression of fibrosis and the development of steatosis. The insulin resistence is frecuently associated with very difficult to cure patients as cirrhotics, afro-american patients, overweight patients and co-infected HCV-HIV patients. Recently is repported that sustained virological (SVR) response in genotype 1 patients is different according the insulin resistance. The SVR was 60% in patients without insulin resistance versus 20% in patients with strong insulin resistance (HOMA > 4.

The present trial desire to analyze the effect that the treatment of insulin resistance produce in higher range of RVS.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with 18 years of age or more
* Serum HCV-RNA quantifiable
* Genotype 1
* Liver disease compensated
* HOMA-IR > 2
* Treatment with Peginterferon alfa-2a + Ribavirin.
* Negative urine or blood pregnancy test (for women of childbearing potential)
* All fertile males and females must be using effective contraception

Exclusion Criteria:

* Liver chirrosis
* Diabetes
* Women with ongoing pregnancy or breast feeding
* HIV positive
* Patients who during 6 months previous to treatment loss more of 10% of weight
* Therapy with anti-neoplasic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 6 months prior to the first dose of study drug
* Any investigational drug 6 weeks prior to the first dose of study drug
* History or other evidence of a medical condition associated with chronic liver disease other than HCV
* Carcinoma hepatocellular
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
* Hgb <12 g/dL in women or <13 g/dL in men or any patient for whom anemia would be medically problematic
* History of significant cardiac disease that could be worsened by acute anemia
* Serum creatinine level >1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Evidence of drug abuse (including excessive alcohol consumption) within one year of study entry
* Inability or unwillingness to provide informed consent or abide by the requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2006-05; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with HCV-RNA | Week 72

SECONDARY OUTCOMES:
Percentage of patients who has erradicated the insulin resistance | week 72

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Romero-Gomez, Dr, Study Director — Hospital Universitario de Valme. Sevilla
Locations (19):
- Spain (19):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital General de Ciudad Real, Ciudad Real, Ciudad Real
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital Clínico Universitario San Cecilio, Granada, Granada
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital de Leon, León, Leon
  - Fundación Hospital de Alcorcón, Alcorcón, Madrid
  - Hospital de la Princesa, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Carlos III, Madrid, Madrid
  - Hospital Puerta de Hierro, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Virgen Macarena, Seville, Sevilla
  - Hospital Universitario de Valme, Seville, Sevilla
  - Hospital General Universitario, Valencia, Valencia